CLINICAL TRIAL: NCT01879345
Title: A Double-blind, Randomized, Placebo-Controlled Study to Evaluate the Tolerability and Pharmacokinetics of Two Single and Multiple High Dose Regimens of BIA 2-093 in Healthy Volunteers
Brief Title: A Study to Evaluate the Tolerability and Pharmacokinetics of Two Single and Multiple High Dose Regimens of BIA 2-093 In Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BIA-2093-113
Record Dates: First submitted 2013-06-13; First posted 2013-06-17 (Estimated); Results first posted 2014-12-30 (Estimated); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: Epilepsy
Keywords: Anticonvulsant
MeSH Terms: conditions — Epilepsy | interventions — eslicarbazepine acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- BIA 2-093 - 1800 mg (Group 1) (Experimental): 3 tablets of BIA 2-093 600 mg
  Interventions: Drug: BIA 2-093 - 1800 mg (Group 1)
- BIA 2-093 - 2400 mg (Group 2) (Experimental): 4 tablets of BIA 2-093 600 mg
  Interventions: Drug: BIA 2-093 - 2400 mg (Group 2)
- Placebo (Placebo Comparator): placebo tablets
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BIA 2-093 - 1800 mg (Group 1) — 3 tablets of BIA 2-093
  Other Names: Eslicarbazepine acetate
  Arms: BIA 2-093 - 1800 mg (Group 1)
Drug: BIA 2-093 - 2400 mg (Group 2) — 4 tablets of BIA 2-093 600 mg
  Other Names: Eslicarbazepine acetate
  Arms: BIA 2-093 - 2400 mg (Group 2)
Drug: Placebo — placebo tablets
  Other Names: sugar pills
  Arms: Placebo

SUMMARY:
Single centre, double-blind, randomised, placebo-controlled study of two dosage regimens of BIA 2-093 - 1800 mg (Group 1) and 2400 mg (Group 2) - in two groups of healthy male volunteers

DETAILED DESCRIPTION:
Within each group (n=9) 3 volunteers were randomised to receive placebo and the remaining 6 volunteers to receive BIA 2-093. No volunteer was a member of more than one treatment group. In each group, the study consisted of a single-dose period (Phase A) followed by a 7-day multiple-dose period (Phase B). The multiple-dose phase started 96 h post single-dose. Progression to the 2400 mg dose (Group 2) only occurred if the 1800 mg dose (Group 1) was considered to be safe and well tolerated. An appropriate interval separated the investigation of the two groups in order to permit a timely review and evaluation of safety data.

Treatment consisted of a single-dose (Phase A) followed by a once-daily dose for 7 days (Phase B). Doses were prepared as follows: Group 1 = 3 tablets of BIA 2-093 600 mg plus 1 placebo tablet, or 4 placebo tablets; Group 2 = 4 tablets of BIA 2-093 600 mg, or 4 placebo tablets.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects aged between 18 and 45 years, inclusive.
* Subjects of body mass index (BMI) between 19 and 30 kg/m2, inclusive.
* Subjects who were healthy as determined by pre-study medical history, physical examination, vital signs, neurological examination, and 12-lead ECG.
* Subjects who had clinical laboratory tests within normal ranges at screening and admission.
* Subjects who had negative tests for HBsAg, anti-HCV Ab and HIV-1 and HIV-2 Ab at screening.
* Subjects who were negative for drugs of abuse and alcohol at screening and admission.
* Subjects who were non-smokers or smoked less than 10 cigarettes or equivalent per day.
* Subjects who were able and willing to give written informed consent.

Exclusion Criteria:

* Subjects who did not conform to the above inclusion criteria, OR
* Subjects who had a clinically relevant history or presence of respiratory, gastrointestinal, renal, hepatic, haematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, endocrine, connective tissue diseases or disorders.
* Subjects who had a clinically relevant surgical history.
* Subjects who had a clinically relevant family history.
* Subjects who had a history of relevant atopy.
* Subjects who had a history of relevant drug hypersensitivity.
* Subjects who had a history of alcoholism or drug abuse.
* Subjects who consumed more than 14 units of alcohol a week.
* Subjects who had a significant infection or known inflammatory process on screening or admission.
* Subjects who had acute gastrointestinal symptoms at the time of screening or admission (e.g., nausea, vomiting, diarrhoea, heartburn).
* Subjects who had used prescription or over-the-counter medication within 2 weeks of admission.
* Subjects who had used any investigational drug or participated in any clinical trial within 3 months of admission.
* Subjects who had previously received BIA 2-093.
* Subjects who had donated or received any blood or blood products within the previous 3 months prior to screening.
* Subjects who were vegetarians, vegans or had medical dietary restrictions.
* Subjects who could not communicate reliably with the investigator.
* Subjects who were unlikely to co-operate with the requirements of the study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2004-10; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Vaz da Silva, MD, PhD, Principal Investigator — Human Pharmacology Unit / BIAL - Portela & Ca, S.A.
Locations (1):
- Human Pharmacology Unit - BIAL - Portela & Ca, S.A., Trofa, Coronado (S.Romão E S. Mamede), Portugal

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: PLC, Placebo
Period: Single-dose Period
Arm/Group | BIA 2-093 - 1800 mg (Group 1) | BIA 2-093 - 2400 mg (Group 2) | Placebo
Started | 6 | 6 | 6
Completed | 6 | 6 | 6
Not Completed | 0 | 0 | 0
Period: 7-day Multiple-dose Period
Arm/Group | BIA 2-093 - 1800 mg (Group 1) | BIA 2-093 - 2400 mg (Group 2) | Placebo
Started | 6 | 6 | 6
Completed | 6 | 6 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BIA 2-093 - 1800 mg (Group 1) | BIA 2-093 - 2400 mg (Group 2) | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 6 | 18
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 6 | 6 | 6 | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events Reported
Description: investigate the tolerability of two single- and multiple-dose regimens of BIA 2-093 (1800 mg and 2400 mg)considering the Number of adverse events reported by patient
Time Frame: 3 weeks
Measure: Number; unit: Number of adverse events reported
Arm/Group | BIA 2-093 - 1800 mg (Group 1) | BIA 2-093 - 2400 mg (Group 2) | Placebo
Number analyzed (Participants) | 6 | 6 | 6
Number of adverse events reported | 10 | 7 | 7

2. Secondary Outcome: Cmax - Maximum Observed Plasma Drug Concentration
Description: Single dose: pharmacokinetic parameters following an oral single-dose of BIA 2-093 Multiple dose: pharmacokinetic parameters following the last dose of an oral 7- day once-daily regimen of BIA 2-093
  Oxcarbazepine is a BIA 2-093 metabolite
Time Frame: Day 1 and Day 7
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- BIA 2-093 - 1800 mg (Group 1): 3 tablets of BIA 2-093 600 mg BIA 2-093 - 1800 mg (Group 1): 3 tablets of BIA 2-093 Oxcarbazepine is a BIA 2-093 metabolite
- BIA 2-093 - 2400 mg (Group 2): 4 tablets of BIA 2-093 600 mg BIA 2-093 - 2400 mg (Group 2): 4 tablets of BIA 2-093 600 mg Oxcarbazepine is a BIA 2-093 metabolite
Arm/Group | BIA 2-093 - 1800 mg (Group 1) | BIA 2-093 - 2400 mg (Group 2)
Number analyzed (Participants) | 6 | 6
ng/mL
  Cmax (BIA 2-005) single dose | 34569 (5623) | 35926 (15301)
  Cmax (BIA 2-005) multiple dose | 47665 (11108) | 56506 (11277)
  Cmax (oxcarbazepine) single dose | 241 (57.1) | 508 (177)
  Cmax (oxcarbazepine) multiple dose | 361 (106) | 734 (186)

3. Secondary Outcome: Tmax - the Time of Occurrence of Cmax
Description: as for outcome 2
Time Frame: Day 1 and Day 7
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | BIA 2-093 - 1800 mg (Group 1) | BIA 2-093 - 2400 mg (Group 2)
Number analyzed (Participants) | 6 | 6
hours
  tmax (BIA 2-005) single dose | 3.8 (1.2) | 3.3 (1.7)
  tmax (BIA 2-005) multiple dose | 2.1 (1.2) | 3.6 (2.7)
  tmax (oxcarbazepine) single dose | 4.67 (1.03) | 4.00 (1.10)
  tmax (oxcarbazepine) multiple dose | 3.83 (1.17) | 3.67 (0.52)

4. Secondary Outcome: AUC0-τ
Description: as for outcome 2
Time Frame: Day 1 and Day 7
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | BIA 2-093 - 1800 mg (Group 1) | BIA 2-093 - 2400 mg (Group 2)
Number analyzed (Participants) | 6 | 6
ng.h/mL
  AUC0-τ (BIA 2-005) single dose | 507563 (86363) | 445596 (116306)
  AUC0-τ (BIA 2-005) multiple dose | 740299 (144882) | 905860 (115783)
  AUC0-τ (oxcarbazepine) single dose | 3589 (847) | 4547 (1512)
  AUC0-τ (oxcarbazepine) multiple dose | 6958 (1824) | 9956 (2329)

ADVERSE EVENTS:
Arm/Group | BIA 2-093 - 1800 mg (Group 1) | BIA 2-093 - 2400 mg (Group 2) | Placebo
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 4/6 | 4/6 | 5/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BIA 2-093 - 1800 mg (Group 1) (N=6) | BIA 2-093 - 2400 mg (Group 2) (N=6) | Placebo (N=6)
Photopsia (Eye disorders) | 0 | 0 | 1
Rhinoconjunctivitis (Eye disorders) | 1 | 0 | 0
Visual disturbance (Eye disorders) | 1 | 0 | 0
Catheter site ecchymosis (Injury, poisoning and procedural complications) | 1 | 0 | 0
Catheter site phlebitis (Injury, poisoning and procedural complications) | 1 | 0 | 0
Blood pressure increased (Investigations) | 0 | 2 | 0
Opticokinetic nystagmus tests abdnormal (Investigations) | 1 | 0 | 1
Knee pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 0 | 0
Paraesthesia circumoral (Nervous system disorders) | 0 | 2 | 0
Pre-syncope (Nervous system disorders) | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 2 | 0
Tremor of hands (Nervous system disorders) | 0 | 0 | 2
Vasovagal reaction (Nervous system disorders) | 0 | 0 | 2
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes